CLINICAL TRIAL: NCT02034812
Title: GenomeDx Decipher Test for Metastatic Disease Prognosis in Prostate Cancer for Patients With Adverse Pathology Post Radical Prostatectomy: Does it Impact Radiation Oncologist' Treatment Recommendations?
Brief Title: Decision Impact Study to Measure the Influence of DECIPHER on Treatment Recommendations for Radiation Oncologists
Acronym: DECIDE3
Status: Completed | Type: Observational
Sponsor: GenomeDx Biosciences Corp (Industry)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CU001.B
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2014-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiation Oncologists: Radiation oncologists targeted for recruitment into the study must meet the following criteria:
  * Practicing, board-certified radiation oncologists
  * Perform consultations on at least 80 patients with prostate cancer annually
  Each participant is asked to complete a questionnaire to assess the impact of Decipher on physicians' treatment recommendation. All participants use the same data collection instrument. Each participant's opinion is collected based on a random selection of cases.
  Interventions: Other: Decipher Questionnaire

INTERVENTIONS:
Other: Decipher Questionnaire — Pathological data from 12 de-identified patient cases will be reviewed by at least 25 Radiation Oncologists before and after exposure to the Decipher test results. Given the number of patient cases, reviewed by each participant, this allows for assessment of decision making based on 300 patient case reviews at each time point, immediately following RP and at the time of PSA rise.

SUMMARY:
This clinical utility study is based on a review of real but de-identified and randomized patient cases and aims to evaluate radiation oncologist's treatment recommendations before and after reviewing the results provided by the Decipher test. The primary intent is to help guide development and design of future clinical utility studies for Decipher.

DETAILED DESCRIPTION:
Patient cases were selected using existing data generated from patient specimens collected in a separate IRB approved protocol, in which pathological specimens were tested to generate a test result for comparison to outcomes. Those test results are presented in this study, but not the individual patient outcomes. Physicians participating in this current study did not provide care for any of the subjects in the previous study. Cases are presented to physicians in a randomized order and in a form that prevents the patients from being identified, directly or indirectly.

High risk patient cases were selected to reflect a range of clinicopathological variables and were further stratified based on the Decipher predicted probability of developing metastasis 5 years after RP and 3 years after BCR (as shown in the table below). High (low) Decipher (GC) risk was defined as a 5- or 3-year predicted probability of metastasis greater (less) than 6% for the adjuvant setting and greater (less) than 18% for the salvage setting.

ELIGIBILITY:
Case Inclusion Criteria:

Patient cases eligible for this study were treated with radical prostatectomy and have one or more adverse pathological features present defined as:

Pathological Gleason score ≥ 8 or Gleason score 7 with primary pattern 4; Pathological stage T3a (= Extracapsular extension) or T3b (=Seminal vesicle invasion); Positive surgical margins Gleason grade upgrade from biopsy to surgery Detectable PSA, defined as failure of PSA to fall to undetectable, or PSA detectable and rising on 2 or more subsequent determinations

Case Exclusion Criteria:

Metastatic disease (M+) prior to surgery Received any neo-adjuvant prostate cancer treatment prior to radical prostatectomy (radiation, hormone, chemotherapy)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians:
  Radiation oncologists targeted for recruitment into the study must meet the following criteria:
  * Practicing, board-certified radiation oncologists.
  * Perform consultations on at least 80 patients with prostate cancer annually.
  Patients:
  Patients diagnosed with localized prostate cancer that received radical prostatectomy as the first line treatment.
  De-identified patient cases were selected from an independent clinical validation study of patients with adverse pathology features treated between 2000 and 2006. (Karnes et al., 2013)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in treatment recommendation | 12 months
  Change in treatment recommendation from pre- to post-Decipher report, defined as any change in treatment recommendation.

SECONDARY OUTCOMES:
Specific change in treatment recommendation | 12 months
  1. Change in treatment recommendation from pre- to post-Decipher report defined as any of the following: Observation to Any treatment Any treatment to Observation
Measure of Intensity of treatment | 12 months
  Change in treatment recommendation from pre- to post-Decipher report involving an increase or decrease in intensity.
Confidence in treatment | 12 months
  Changes in Radiation Oncologist's expressed level of confidence in the treatment recommendation
Utility of Decipher test | 12 months
  Radiation Oncologist's perception regarding the utility of the Decipher test

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Nguyen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Cooperberg MR, Hilton JF, Carroll PR. The CAPRA-S score: A straightforward tool for improved prediction of outcomes after radical prostatectomy. Cancer. 2011 Nov 15;117(22):5039-46. doi: 10.1002/cncr.26169. Epub 2011 Jun 3. PMID 21647869
- [Background] Pound CR, Partin AW, Eisenberger MA, Chan DW, Pearson JD, Walsh PC. Natural history of progression after PSA elevation following radical prostatectomy. JAMA. 1999 May 5;281(17):1591-7. doi: 10.1001/jama.281.17.1591. PMID 10235151
- [Background] Bolla M, van Poppel H, Collette L, van Cangh P, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Marechal JM, Scalliet P, Haustermans K, Pierart M; European Organization for Research and Treatment of Cancer. Postoperative radiotherapy after radical prostatectomy: a randomised controlled trial (EORTC trial 22911). Lancet. 2005 Aug 13-19;366(9485):572-8. doi: 10.1016/S0140-6736(05)67101-2. PMID 16099293
- [Background] Thompson IM Jr, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathologically advanced prostate cancer: a randomized clinical trial. JAMA. 2006 Nov 15;296(19):2329-35. doi: 10.1001/jama.296.19.2329. PMID 17105795
- [Background] Wiegel T, Bottke D, Steiner U, Siegmann A, Golz R, Storkel S, Willich N, Semjonow A, Souchon R, Stockle M, Rube C, Weissbach L, Althaus P, Rebmann U, Kalble T, Feldmann HJ, Wirth M, Hinke A, Hinkelbein W, Miller K. Phase III postoperative adjuvant radiotherapy after radical prostatectomy compared with radical prostatectomy alone in pT3 prostate cancer with postoperative undetectable prostate-specific antigen: ARO 96-02/AUO AP 09/95. J Clin Oncol. 2009 Jun 20;27(18):2924-30. doi: 10.1200/JCO.2008.18.9563. Epub 2009 May 11. PMID 19433689
- [Background] Thompson IM, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathological T3N0M0 prostate cancer significantly reduces risk of metastases and improves survival: long-term followup of a randomized clinical trial. J Urol. 2009 Mar;181(3):956-62. doi: 10.1016/j.juro.2008.11.032. Epub 2009 Jan 23. PMID 19167731
- [Background] Schreiber D, Rineer J, Sura S, Teper E, Nabhani T, Han P, Schwartz D, Choi K, Rotman M. Radical prostatectomy for cT3-4 disease: an evaluation of the pathological outcomes and patterns of care for adjuvant radiation in a national cohort. BJU Int. 2011 Aug;108(3):360-5. doi: 10.1111/j.1464-410X.2010.09875.x. Epub 2010 Nov 18. PMID 21087395
- [Background] Krupski TL, Foley KA, Baser O, Long S, Macarios D, Litwin MS. Health care cost associated with prostate cancer, androgen deprivation therapy and bone complications. J Urol. 2007 Oct;178(4 Pt 1):1423-8. doi: 10.1016/j.juro.2007.05.135. Epub 2007 Aug 16. PMID 17706711
- [Background] Ross AE, Feng FY, Ghadessi M, Erho N, Crisan A, Buerki C, Sundi D, Mitra AP, Vergara IA, Thompson DJ, Triche TJ, Davicioni E, Bergstralh EJ, Jenkins RB, Karnes RJ, Schaeffer EM. A genomic classifier predicting metastatic disease progression in men with biochemical recurrence after prostatectomy. Prostate Cancer Prostatic Dis. 2014 Mar;17(1):64-9. doi: 10.1038/pcan.2013.49. Epub 2013 Oct 22. PMID 24145624
- [Background] Erho N, Crisan A, Vergara IA, Mitra AP, Ghadessi M, Buerki C, Bergstralh EJ, Kollmeyer T, Fink S, Haddad Z, Zimmermann B, Sierocinski T, Ballman KV, Triche TJ, Black PC, Karnes RJ, Klee G, Davicioni E, Jenkins RB. Discovery and validation of a prostate cancer genomic classifier that predicts early metastasis following radical prostatectomy. PLoS One. 2013 Jun 24;8(6):e66855. doi: 10.1371/journal.pone.0066855. Print 2013. PMID 23826159
- [Background] Karnes RJ, Bergstralh EJ, Davicioni E, Ghadessi M, Buerki C, Mitra AP, Crisan A, Erho N, Vergara IA, Lam LL, Carlson R, Thompson DJ, Haddad Z, Zimmermann B, Sierocinski T, Triche TJ, Kollmeyer T, Ballman KV, Black PC, Klee GG, Jenkins RB. Validation of a genomic classifier that predicts metastasis following radical prostatectomy in an at risk patient population. J Urol. 2013 Dec;190(6):2047-53. doi: 10.1016/j.juro.2013.06.017. Epub 2013 Jun 11. PMID 23770138
- [Background] Badani K, Thompson DJ, Buerki C, Davicioni E, Garrison J, Ghadessi M, Mitra AP, Wood PJ, Hornberger J. Impact of a genomic classifier of metastatic risk on postoperative treatment recommendations for prostate cancer patients: a report from the DECIDE study group. Oncotarget. 2013 Apr;4(4):600-9. doi: 10.18632/oncotarget.918. PMID 23592338
- [Background] Erho N, Buerki C, Triche TJ, Davicioni E, Vergara IA. Transcriptome-wide detection of differentially expressed coding and non-coding transcripts and their clinical significance in prostate cancer. J Oncol. 2012;2012:541353. doi: 10.1155/2012/541353. Epub 2012 Aug 16. PMID 22956952